CLINICAL TRIAL: NCT04019548
Title: Patient Reported Outcomes in Term of Swallowing and Quality of Life After Prophylactic Versus Reactive Percutaneous Endoscopic Gastrostomy Tube Placement in Advanced Oropharyngeal Cancer Patients Treated With Definitive Chemo-radiotherapy
Brief Title: Assessment of Swallowing Function and Quality of Life in Oropharyngeal Cancer Patients Treated by Chemo-radiotherapy
Acronym: SwallPEG
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IJB-RT-HNC-001
Record Dates: First submitted 2019-05-10; First posted 2019-07-15 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Oropharyngeal Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Cisplatin; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Open-label, randomized study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic PEG (Experimental): Prophylactic PEG tube will be placed before the start of the study treatment (CRT). The enteral nutrition will start following the assessment by the clinical dietitian in order to complete the current oral consumption according to the estimated energy needs (on the basis of 30 to 35 kcal / kg adapted and 1.2 to 1.5 g / prot./ kg.BW) with an increase as needed during the treatment.
  Interventions: Device: Percutaneous Endoscopic Gastrotomy tube placement; Drug: Cisplatin injection; Radiation: Radiotherapy
- Reactive PEG (Experimental): Reactive PEG tube will be placed and enteral nutrition initiated, during the study treatment period in case of decrease of oral intake less than 2/3 of estimated energy requirements (based on 30-35 kcal / adapted kg .BW and 1.2 - 1.5 g/prot./adapted kg. BW) for a period of or anticipated to be, greater than 7 days or weight loss ≥ 5% from pre-treatment baseline).
  Interventions: Device: Percutaneous Endoscopic Gastrotomy tube placement; Drug: Cisplatin injection; Radiation: Radiotherapy

INTERVENTIONS:
Device: Percutaneous Endoscopic Gastrotomy tube placement — placement of the PEG tube depends on arm
Drug: Cisplatin injection — Two therapeutic regimen allowed:
  * Days 1 and 22 : cisplatin 100mg/m2 IV
  * Days 1,8,15,22,29,36: weekly cisplatin 40 mg/m2 IV
Radiation: Radiotherapy — Simultaneous integrated boost (SIB) intensity modulated radiotherapy (IMRT). The median dose prescription will be 32 x 2.16 Gy to the high risk PTV and 32 x 1.75 Gy to the elective PTV.

SUMMARY:
Open-label, interventional, multicentric, randomized, phase III study. Cancer studied is the oropharyngeal cancer.

Study is composed by 2 arms of subjects: prophylactic or reactive percutaneous endoscopic gastrostomy tube placement.

All subjects will be treated with a cisplatin standard chemotherapy regimen and by simultaneous integrated boost (SIB) intensity modulated radiotherapy (IMRT).

DETAILED DESCRIPTION:
Open-label, interventional, multicentric, randomized, phase III study. Cancer studied is the oropharyngeal cancer.

Study is composed by 2 arms of subjects (male or female): prophylactic or reactive percutaneous endoscopic gastrostomy tube placement.

The arm will be allocated by randomisation (1:1).

* Prophylactic PEG (pPEG): Prophylactic PEG tube will be placed before the start of the study treatment (CRT). The enteral nutrition will start following the assessment by the clinical dietitian in order to complete the current oral consumption according to the estimated energy needs (on the basis of 30 to 35 kcal / kg adapted and 1.2 to 1.5 g / prot./ kg.BW) with an increase as needed during the treatment.
* Reactive PEG (rPEG): Reactive PEG tube will be placed and enteral nutrition initiated, during the study treatment period in case of decrease of oral intake less than 2/3 of estimated energy requirements (based on 30-35 kcal / adapted kg .BW and 1.2 - 1.5 g/prot./adapted kg. BW) for a period of or anticipated to be, greater than 7 days or weight loss ≥ 5% from pre-treatment baseline).

All subjects will be treated with a cisplatin standard chemotherapy regimen and by simultaneous integrated boost (SIB) intensity modulated radiotherapy (IMRT).

Cisplatin: Two therapeutic regimens are allowed:

* Days 1 and 22: cisplatin 100mg/m2 IV
* Days 1,8,15,22,29 and 39: weekly cisplatin 40mg/m2 IV

Radiotherapy: The median dose prescription will be 32 x 2.16 Gy to the high risk PTV and 32 x 1.75 Gy to the elective PTV.

Medical device: The medical device used in this trial is a percutaneous endoscopic gastrostomy tube with the CE label: CE0120. The medical device is used in the indication of the notice.

The estimated number of subjects to screen is 121 patients for an estimated number of 110 patients randomised for 100 evaluable patients.

The end of study will be declared when all the following criteria will have been met:

* The study ends after last visit of the last patient remaining in the study.
* The trial is mature for the analysis of the endpoints as defined in the protocol, if the trial reaches its endpoints.
* The database has been fully cleaned and frozen for all analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. ECOG performance status ≤ 2
3. Female and Male
4. Newly diagnosed, histologically confirmed primary squamous cell carcinoma of the oropharynx
5. Candidate for curative intent radiotherapy and systemic treatment
6. No prior or current anticancer treatment for the HNSCC (e.g. neo-adjuvant chemotherapy, surgery)
7. Diagnosis biopsy results
8. HPV/p 16 testing results
9. Serum test (for subjects of childbearing potential) negative within 7 days prior to the 1st CRT administration.
10. Women of childbearing potential must agree to use of one highly effective method of contraception prior study entry, during the course of the study and at least 6 months after the last administration of cisplatin.
11. Men with childbearing potential partner must agree to use condom during the course of this study and for at least 6 months after the last administration of the cisplatin.
12. Adequate bone marrow function as defined below:

    * Absolute neutrophil count (ANC) ≥1500/µL or 1.5x109/L
    * Hemoglobin ≥ 9 g/dL
    * Platelets ≥100000/µL or 100x109/L
13. Adequate liver function as defined below:

    * Serum total bilirubin ≤ 1.5 x ULN. In case of known Gilbert's syndrome < 3 x UNL is allowed
    * AST (SGOT)/ALT (SGPT) ≤ 2.5 x ULN
    * Alkaline phosphatase ≤ 2.5 x ULN
14. Adequate renal function as defined below:

    * Creatinine ≤ 1.5 x UNL and creatinine clearance > 60 mL/min
15. Peripheral neuropathy ≤ grade 1
16. Hear impaired ≤ grade 1
17. Completion of all necessary screening procedures within 15 days prior to randomisation.
18. Signed Informed Consent form (ICF) obtained prior to any study related procedure.
19. Ability to understand and complete the questionnaires (language proficiency, cognitive functioning) as judged by principal investigator upon screening

Exclusion Criteria:

1. Severe malnutrition
2. Dysphagia requiring a liquid or puree texture modified diet (grade ≥ 2 (CTCAE_v.5)
3. Distant metastasis
4. Serious coagulation disorders (INR>1.5, PTT>50s, platelets <50000/mm3)
5. Subject with a significant medical, neuro-psychiatric, or surgical condition, currently uncontrolled by treatment, which, in the principal investigator's opinion, may interfere with completion of the study.
6. Other malignancies in the 3 years prior to study entry except of surgically cured carcinoma in situ of the cervix, in situ breast cancer, incidental finding of stage T1a or T1b prostate cancer, and basal/squamous cell carcinoma of the skin;
7. Pregnant and/or lactating women.
8. Known hypersensitivity to the study drug (cisplatin) or excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
global M.D. Anderson Dysphagia Inventory score at 6 months after end of treatment. | at 6 months after end of treatment
  The M.D.Anderson Dysphagia inventory is a dysphagia-specific quality-of-life questionnaire for patients with H&N cancer including 20 items divided into 4 subscales emotional (6 questions), functional (5 questions), physical (8 questions) and one global question. Each subscale has a score ranging from 1 to 5 (higher scores represent a better outcome). The mean score of the 20 items will be multiplied by a factor of 20 to obtain a MDADI total score which ranges from 20 (extremely low functioning) to 100 (high functioning). A difference of 8 points in MDADI score is considered as the Minimal Clinically Important Difference for the trial.

SECONDARY OUTCOMES:
Assessment of Quality of Life | Baseline; at week 3 & 6 during treatment; at 1,3, 6, 12 and 24 months after end of treatment
  Outcome measure: completion of EORTC QLQ-C30 questionnaire
Assessment of Quality of Life | Baseline; at week 3 & 6 during treatment; at 1,3, 6, 12 and 24 months after end of treatment
  Outcome measure: completion of EORTC QLQ-H&N43 module questionnaire
Assessment of Quality of Life | Baseline; at week 3 & 6 during treatment; at 1,3, 6, 12 and 24 months after end of treatment
  Outcome measure: completion of FACT-HN questionnaire
Assessment of chemo-radiotherapy treatment related toxicities and PEG tube placement complications | through study completion, an average of 38 months
  Outcome measure: Incidence, type and severity of all adverse events (AEs) and serious adverse events according to CTCAE version 5.0 ;
Assessment of chemo-radiotherapy treatment related toxicities and PEG tube placement complications | through study completion, an average of 38 months
  Outcome measure:Incidence, type and severity of radiotherapy related AEs also according to Radiation Therapy Oncology Group (RTOG) / European Organisation for Research and treatment of Cancer (EORTC) scores; In the RTOG/EORTC Late Radiation Morbidity Scoring, 0 means an absence of radiation effects and 5 means the effects led to death. The severity of reactions is graded from 1 through 4.
Assessment of chemo-radiotherapy treatment related toxicities and PEG tube placement complications | through study completion, an average of 38 months
  Outcome measure:Severity of oropharyngeal mucositis and swallowing disorders according to Internal consensus scale (ICS);
Assessment of chemo-radiotherapy treatment related toxicities and PEG tube placement complications | through study completion, an average of 38 months
  Outcome measure: Oropharyngeal mucositis according to the oral mucositis weekly questionnaire-Head and Neck cancer (OMWQ-NH) completed by the subject;
Assessment of chemo-radiotherapy treatment related toxicities and PEG tube placement complications | through study completion, an average of 38 months
  Outcome measure: Salivary toxicity according to the xerostomia questionnaire completed by the subject.
Impact of the nutritional status on survival and toxicity outcomes | Baseline, during treatment period (7 weeks) and follow-up period (24 months)
  Outcome measure: Clinical dietitian assessment including risk screening by Nutritional Risk Screening 2002 (NRS-2002)
Impact of the nutritional status on survival and toxicity outcomes | Baseline, during treatment period (7 weeks) and follow-up period (24 months)
  Outcome measure: Clinical dietitian assessment using GLIM criteria (Global Leadership Initiative on Malnutrition criteria).
Assessment of clinical tumour response after study treatment | at 3 and 12 months after end of treatment
  Outcome measure:Tumour response after study treatment measured by DECT and PET-CT
Assessment of the subject outcome | at 3, 12 and 36 months after end of treatment
  Outcome measure: loco regional control (LRC)
Assessment of the subject outcome | at 3, 12 and 36 months after end of treatment
  Outcome measure: distant recurrence/distant progression (DR/DP)
Assessment of the subject outcome | at 3, 12 and 36 months after end of treatment
  Outcome measure: second primary (SP)
Assessment of the subject outcome | at 3, 12 and 36 months after end of treatment
  Outcome measure: disease-free survival (DFS)
Assessment of the subject outcome | at 3, 12 and 36 months after end of treatment
  Outcome measure: disease specific survival (DSS)
Assessment of the subject outcome | at 3, 12 and 36 months after end of treatment
  Outcome measure: overall survival (OS)
Impact of tobacco consumption on the outcomes | Baseline, at week 3 and at 1, 3, 6, 12 and 24 months after the end of treatment.
  Outcome measure: Assessment of the smoking consumption
Impact of HPV on the outcomes | at screening
  Outcome measure: HPV/p16 status
Cost-Effectiveness of each treatment strategy | during the pre-study treatment period (within 15 days after randomisation and before starting study treatment) and at 12 months after end of treatment
  Outcome measure: EuroQol 5D5L Questionnaire
Clinical validation of cancer prediction models available at www.predictcancer.org | at 6 months after treatment
  HPV-based prognostic nomogram for oro-pharyngeal carcinoma
Clinical validation of cancer prediction models available at www.predictcancer.org | at 6 months after treatment
  prediction tool for swallowing dysfunction, xerostomia, sticky saliva and tube feeding dependence

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - CHU Saint Pierre, Brussels
  - Institut Jules Bordet, Brussels

REFERENCES:
- [Derived] Dragan T, Van Gossum A, Duprez F, Lalami Y, Lefebvre Y, Mootassim-Billah S, Beauvois S, Gulyban A, Vandekerkhove C, Boegner P, Paesmans M, Ameye L, Digonnet A, Quiriny M, Dequanter D, Lipski S, Willemse E, Rodriguez A, Carlot S, Karaca Y, Lemort M, Emonts P, Al Wardi C, Van Gestel D. Patient-reported outcomes in terms of swallowing and quality of life after prophylactic versus reactive percutaneous endoscopic gastrostomy tube placement in advanced oropharyngeal cancer patients treated with definitive chemo-radiotherapy: Swall PEG study. Trials. 2022 Dec 21;23(1):1036. doi: 10.1186/s13063-022-06991-6. PMID 36539781